CLINICAL TRIAL: NCT06237647
Title: Comparison of Steroid, Platelet-rich Plasma and Platelet-rich Plasma Plus Hyaluronic Acid Injection for Rotator Cuff Lesions
Brief Title: Comparison of Steroid, PRP,and PRP Plus Hyaluronic Acid Injection for Rotator Cuff Lesions.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tien-Ching Lee (Other)
Responsible Party: Sponsor-Investigator, Tien-Ching Lee, Department of Orthopaedics, Kaohsiung Medical University
Organization: Kaohsiung Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT-002
Record Dates: First submitted 2023-12-20; First posted 2024-02-01 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Rotator Cuff Lesions
Keywords: rotator cuff lesions
MeSH Terms: interventions — Hyaluronic Acid; Glucose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PRP+HA (Experimental): 5mL of PRP+HA
  Interventions: Dietary Supplement: Hyaluronic acid, HA
- PRP injection (No Intervention): 4mL of PRP added 1 mL of lidocaine
- Steroid (No Intervention): 1 mL of rinderon added 4 mL of lidocaine
- PROLOTHERAPHY (Experimental): 4 mL of 20% dextrose added1 mL lidocaine
  Interventions: Dietary Supplement: Hyaluronic acid, HA

INTERVENTIONS:
Dietary Supplement: Hyaluronic acid, HA — improve tissue repair
  Other Names: glucose
  Arms: PROLOTHERAPHY; PRP+HA

SUMMARY:
Rotator cuff tear is a common cause of shoulder pain. Steroids, hyaluronic acid (HA), and platelet-rich plasma (PRP) injections are becoming popular for the treatment of chronic rotator cuff partial tear. The investigators plan to evaluate the effect of the new product of PRP combined with HA on the rotator cuff and prove its benefit of pain control and function recovery.

DETAILED DESCRIPTION:
Rotator cuff tear is a common cause of shoulder pain. Steroids, hyaluronic acid (HA), and platelet-rich plasma (PRP) injections are becoming popular for the treatment of chronic rotator cuff partial tear. The investigators plan to evaluate the effect of the new product of PRP combined with HA on the rotator cuff and prove its benefit of pain control and function recovery.

1. Name: Cellular matrix™ PRP-HA
2. Dosage form: Cellular Matrix A-CP-HA Kit (Ref. A-CP-HA-3)
3. Dose(s): 3 mL of platelet-rich plasma (PRP) combined with 2 mL of hyaluronic acid
4. Dosing schedule: one injection. After collecting 6 mL of blood collection and then centrifugation for 5 minutes, the PRP with a platelet concentration 1.5-1.6 times higher than the baseline in blood, deprived of contamination with red and white blood cells, entrapped in a 3D network of HA
5. Mechanism of action: PRP contains rich growth factors and HA could function as bio-scaffold. They have a synergic effect on tissue repair.
6. Pharmacological category: class III medical device

ELIGIBILITY:
Inclusion Criteria:

* A. Shoulder pain for at least 1 months
* B.partial-thickness tear diagnosed by MRI or Echo
* C.age between 20 and 85 years old

Exclusion Criteria:

* A. inflammatory disease, such as rheumatoid arthritis, SLE, etc.
* B. pregnancy
* C. known malignancy
* D. hematologic disease (or hemoglobin <10 g/dl, platelet <150.000 ul)
* E. history of shoulder infection
* F. history of shoulder surgery
* G. prior steroid injection for 3 times or more
* H. full-thickness tear
* I. other shoulder problems, such as osteoarthritis, fracture malunion, etc.
* J. subjects who cannot comply with the protocol of study
* K. The shoulder pain area has been treated with PRP for less than 3 months

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Constant-Murley Shoulder Score (CMSS) | before treatment, 4-week, 12-week, 24-week.
  The Constant-Murley Shoulder Score (CMSS) is a multi-item functional scale assessing pain, ADL, ROM, and strength of the affected shoulder. score: 0-100. The higher score means the function feels good and painless.

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) Score | before treatment, 4-week, 12-week, 24-week.
  The American Shoulder and Elbow Surgeons Shoulder Score (ASES) was created by the Society of the American Shoulder and Elbow Surgeons in 1994 as a tool that applies to all shoulder diagnoses. score: 0-100. The higher score means the function feels good and painless.
range of motion of shoulder | before treatment, 4-week, 12-week, 24-week.
  ROM: flex, extension, abduction, adduction, internal rotation, external rotation. degree: 0-180. The higher degree means the shoulder rotation extends good and is painless.
pain score (VAS) | before treatment, 4-week, 12-week, 24-week.
  score 0-10. The lower score means the function feels good and painless.
the change of anatomy | before treatment, 4-week, 12-week, 24-week.
  Echo or MRI_Measure the wound size of rotator muscle rupture and confirm whether the wound has healed
associated complications | before treatment, 4-week, 12-week, 24-week.
  infection, surgery, hypertrophic scar, consistent pain, etc. After the trial, the investigators calculate the rate of these complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Sanmin, Taiwan

DOCUMENTS (1):
  • Informed Consent Form (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT06237647/ICF_000.pdf